CLINICAL TRIAL: NCT04610515
Title: Innovative Support for Patients With SARS-COV2 Infections (COVID-19) Registry (INSPIRE)
Acronym: INSPIRE
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Collaborators: Yale University (Other); University of Washington (Other); Thomas Jefferson University (Other); University of California, Los Angeles (Other); University of California, San Francisco (Other); University of Texas Southwestern Medical Center (Other); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Michael Gottlieb, Associate Professor of Emergency Medicine, Rush University Medical Center
Other Study IDs: 75D30120C08008
Record Dates: First submitted 2020-10-28; First posted 2020-10-30 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-07

CONDITIONS: Covid19; ME/CFS; SARS COV2; Novel Coronavirus Infection; Neurocognitive Disorders; Cardiovascular Diseases
MeSH Terms: conditions — COVID-19; Fatigue Syndrome, Chronic; Neurocognitive Disorders; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Symptomatic Individuals with infection with SARS-COV2 (ie exposed cohort): Symptomatic Individuals test positive for SARS-COV2. Participants will be enrolled soon after infection and followed to assess for long term outcomes.
- Symptomatic Individuals without infection with SARS-COV2 (ie unexposed cohort): Symptomatic Individuals test negative for SARS-COV2. Participants will be enrolled soon after testing and followed to assess for long term outcomes.

SUMMARY:
The Innovative Support for Patients with SARS COV-2 Infections Registry (INSPIRE) study is a CDC-funded COVID-19 project to understand the long-term health outcomes in recently tested adults, both negative and positive, who have suspected COVID symptoms at the time of their test. Participants will complete short online surveys every 3 months for 18 months, share information about their health using a secure web-based platform, and are compensated for their time.

DETAILED DESCRIPTION:
This study will use a digital platform to longitudinally track comprehensive information including patient self-report as well as data that describe the process and outcome of care in the electronic medical record (EMR) of a large representative sample of patients under investigation for SARSCOV2. The objective is to generate knowledge rapidly using digital tools and collaborative sciences to produce real-time data, analysis, and reporting compared to more traditional approaches. An additional goal is to promote an open science approach whereby scientists, with proper approvals and in line with the permissions granted by the participants, have the opportunity to work with data in ways that protect individual privacy but promote rapid dissemination and implementation of knowledge.

ELIGIBILITY:
INCLUSION CRITERIA

1. Fluent in English or Spanish;
2. Age 18 and over;
3. Self-reported symptoms suggestive of acute SARSCOV2 infection;
4. Under investigation for SARSCOV2 (defined as a patient who has received any screening or diagnostic test used to detect the presence of COVID19 including any FDA approved or authorized molecular or antigen-based assay) within the last 42 days.

EXCLUSION CRITERIA

1. Unable to provide informed consent;
2. Study team unable to confirm result of diagnostic test for SARSCOV2;
3. Does not have access to a hand-held device or computer that would allow for digital participation in the study;
4. Individuals who are prisoners while participating in the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults aged>=18, with symptoms consistent with infection with SARS-COV2; test positive vs test negative individuals will be enrolled at a rate of 3:1.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Assess for medium and long-term sequalae of SARS-CoV-2 infection | 18 months post enrollment
  Clinical phenotypes of sequelae will be determined at the time of analysis based on published literature

SECONDARY OUTCOMES:
Incident myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS) | 18 months post enrollment
  Determine the risk of myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS) in those with symptoms of SARSCOV2 infection with vs. without a positive confirmatory test.
Ambulatory care and/or ED visits post enrollment | 18 months post enrollment
  Count of ambulatory care and/or ED visits post enrollment as obtained from the EMR
Hospitalizations post enrollment | 18 months post enrollment
  Count of hospitalizations post enrollment as obtained from the EMR
Death during hospital admission | 18 months post enrollment
  Death during hospital admission as determined by data from the EMR
Hospital-free survival | 18 months post enrollment
  Hospital-free survival as determined by data from the EMR
ICU-free survival | 18 months post enrollment
  ICU-free survival as determined by data from the EMR

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gottlieb, MD, Principal Investigator — Rush University Medical Center; Robert A Weinstein, MD, Principal Investigator — Rush University Medical Center
Locations (8):
- United States (8):
  - UCLA, Los Angeles, California
  - UCSF, San Francisco, California
  - Yale, New Haven, Connecticut
  - Rush University Medical Center, Chicago, Illinois
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wisk LE, Gottlieb M, Chen P, Yu H, O'Laughlin KN, Stephens KA, Nichol G, Montoy JCC, Rodriguez RM, Santangelo M, Gatling K, Spatz ES, Venkatesh AK, Rising KL, Hill MJ, Huebinger R, Idris AH, Willis M, Kean E, McDonald SA, Elmore JG, Weinstein RA. Association of SARS-CoV-2 With Health-related Quality of Life 1 Year After Illness Using Latent Transition Analysis. Open Forum Infect Dis. 2025 Jun 10;12(6):ofaf278. doi: 10.1093/ofid/ofaf278. eCollection 2025 Jun. PMID 40496983
- [Derived] Hill MJ, Huebinger RM, Ebna Mannan I, Yu H, Wisk LE, O'Laughlin KN, Gentile NL, Stephens KA, Gottlieb M, Weinstein RA, Koo K, Santangelo M, Saydah S, Spatz ES, Lin Z, Schaeffer K, Kean E, Montoy JCC, Rodriguez RM, Idris AH, McDonald S, Elmore JG, Venkatesh A. Race, Ethnicity, and Gender Differences in Patient Reported Well-Being and Cognitive Functioning Within 3 Months of Symptomatic Illness During COVID-19 Pandemic. J Racial Ethn Health Disparities. 2025 Oct;12(5):3192-3209. doi: 10.1007/s40615-024-02124-8. Epub 2024 Aug 22. PMID 39172356
- [Derived] Gottlieb M, Spatz ES, Yu H, Wisk LE, Elmore JG, Gentile NL, Hill M, Huebinger RM, Idris AH, Kean ER, Koo K, Li SX, McDonald S, Montoy JCC, Nichol G, O'Laughlin KN, Plumb ID, Rising KL, Santangelo M, Saydah S, Wang RC, Venkatesh A, Stephens KA, Weinstein RA; INSPIRE Group. Long COVID Clinical Phenotypes up to 6 Months After Infection Identified by Latent Class Analysis of Self-Reported Symptoms. Open Forum Infect Dis. 2023 May 31;10(7):ofad277. doi: 10.1093/ofid/ofad277. eCollection 2023 Jul. PMID 37426952
- [Derived] Wang RC, Gottlieb M, Montoy JCC, Rodriguez RM, Yu H, Spatz ES, Chandler CW, Elmore JG, Hannikainen PA, Chang AM, Hill M, Huebinger RM, Idris AH, Koo K, Li SX, McDonald S, Nichol G, O'Laughlin KN, Plumb ID, Santangelo M, Saydah S, Stephens KA, Venkatesh AK, Weinstein RA; Innovative Support for Patients with SARS-CoV-2 Infections Registry (INSPIRE) Group. Association Between SARS-CoV-2 Variants and Frequency of Acute Symptoms: Analysis of a Multi-institutional Prospective Cohort Study-December 20, 2020-June 20, 2022. Open Forum Infect Dis. 2023 May 23;10(7):ofad275. doi: 10.1093/ofid/ofad275. eCollection 2023 Jul. PMID 37426947
- [Derived] Gottlieb M, Wang RC, Yu H, Spatz ES, Montoy JCC, Rodriguez RM, Chang AM, Elmore JG, Hannikainen PA, Hill M, Huebinger RM, Idris AH, Lin Z, Koo K, McDonald S, O'Laughlin KN, Plumb ID, Santangelo M, Saydah S, Willis M, Wisk LE, Venkatesh A, Stephens KA, Weinstein RA; Innovative Support for Patients with SARS-CoV-2 Infections Registry (INSPIRE) Group. Severe Fatigue and Persistent Symptoms at 3 Months Following Severe Acute Respiratory Syndrome Coronavirus 2 Infections During the Pre-Delta, Delta, and Omicron Time Periods: A Multicenter Prospective Cohort Study. Clin Infect Dis. 2023 Jun 8;76(11):1930-1941. doi: 10.1093/cid/ciad045. PMID 36705268
- [Derived] Spatz ES, Gottlieb M, Wisk LE, Anderson J, Chang AM, Gentile NL, Hill MJ, Huebinger RM, Idris AH, Kinsman J, Koo K, Li SX, McDonald S, Plumb ID, Rodriguez RM, Saydah S, Slovis B, Stephens KA, Unger ER, Wang RC, Yu H, Hota B, Elmore JG, Weinstein RA, Venkatesh A. Three-Month Symptom Profiles Among Symptomatic Adults With Positive and Negative Severe Acute Respiratory Syndrome Coronavirus 2 Tests: A Prospective Cohort Study From the INSPIRE Group. Clin Infect Dis. 2023 May 3;76(9):1559-1566. doi: 10.1093/cid/ciac966. PMID 36573005